CLINICAL TRIAL: NCT05423873
Title: A Multi-Center Clinical Trial to Evaluate the Efficacy and Tolerability for Treatment of Facial Hyperpigmentation and Photodamaged Skin With a Dual Regimen Treatment Containing Vitamin C and a Tinted SPF 45 Moisturizer
Brief Title: A Multi-Center, Open-label Study Evaluate the Efficacy and Tolerability of a Dual Skincare Regimen Treatment for Facial Hyperpigmentation and Photodamaged Skin in Patients Exposed to Extrinsic Factors of Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Revision Skincare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RS-2020-04
Record Dates: First submitted 2022-06-13; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Hyperpigmentation; Photodamaged Skin; Wrinkle; Fine Lines
Keywords: Vitamin C; Sunscreen; Pollution; Solar Radiation
MeSH Terms: conditions — Hyperpigmentation

STUDY DESIGN:
Intervention Model Description: Prospective, Multi-Center, Open-Label 33 female subjects between 35 to 60 years old with Fitzpatrick skin type I-V, moderate to severe global face hyperpigmentation, and moderate global face photodamage.
  Washout period of 2 weeks refraining from active antiaging topical products, including vitamin C, retinoids, peptides, and growth factors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin C Serum and Moisturizing Sunscreen SPF 45 (Other): Dual Regimen:
  Vitamin C Serum Tinted Moisturizing Sunscreen SPF 45
  Interventions: Other: Gentle Cleansing Lotion, Revision Skincare

INTERVENTIONS:
Other: Gentle Cleansing Lotion, Revision Skincare — Gentle cleansing lotion to be used by study participants twice daily

SUMMARY:
This open-label, multi-center clinical trial was conducted to evaluate the dual skincare regimen of vitamin C serum and moisturizing sunscreen SPF 45 to improve facial hyperpigmentation and photodamage after 12 weeks of twice daily use in healthy female subjects between 35 - 60 years old. A total of 33 subjects completed study participation.

DETAILED DESCRIPTION:
This open-label, multi-center clinical trial was conducted to evaluate the dual skincare regimen of vitamin C serum and moisturizing sunscreen SPF 45 to improve facial hyperpigmentation and photodamage when used twice daily over the course of 12 weeks by healthy women with Fitzpatrick skin type I - V, moderate to severe global face hyperpigmentation and moderate global face photodamage.

Efficacy and tolerability will be assessed through clinical grading at baseline, weeks 4, 8 and 12. Efficacy evaluation for hyperpigmentation (mottled), hyperpigmentation (discrete), overall photodamage, clarity/brightness, overall appearance, skin tone evenness (redness), fine lines and wrinkles. Investigator and subject tolerability, self-assessment questionnaire and clinical VISIA photography will be completed at baseline, weeks 4, 8 and 12. Subject testimonials will be completed at week 12.

A total of 33 subjects completed study participation.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 35 and 60 years old.
* Women with Fitzpatrick skin type I-V.
* Subjects must have moderate to severe global face hyperpigmentation.
* Subjects must have moderate global face photodamage.
* Subjects must have no known medical conditions that, in the investigator's opinion, may interfere with study participation.
* Subjects must be willing to provide verbal understanding and written informed consent.

Exclusion Criteria:

* Subjects which had a health condition and/or pre-existent dormant dermatological disease on the face.
* Subjects that are unwilling to comply with the protocol.
* Female subjects who are pregnant, breast feeding, or planning a pregnancy.
* Subjects who have demonstrated a previous hypersensitivity reaction to any of the ingredients of the study products.
* Subjects who have a history of skin cancer.
* Subjects who have observable suntan, sunburn, scars, nevi, tattoo, excess hair, etc. or other dermatological condition on the face that might influence the test results in the opinion of the investigator.
* Subjects who have routinely used any anti-aging, anti-wrinkles, antioxidants treatments and skin-firming products less than 30 days prior to the study entry.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Improvement in clinical efficacy of hyperpigmentation versus Baseline | 12 weeks
  The primary efficacy endpoint will be the Investigator Clinical Grading using Modified Griffith's 10-point Scale. A change in scores at week 4, week 8 and week 12 in comparison to baseline indicates an improvement for the indicated parameter.
  Global facial hyperpigmentation will be assessed on each subject's face using a modified Griffiths' 10-point scale according to the following numerical definitions (half-point scores may be used as necessary to more accurately describe the skin condition): 0 = none (best possible condition); 1 to 3 = mild; 4 to 6 = moderate;7 to 9 = severe (worst possible condition). The lower the score equates to the best possible outcome.
Lack of Significant Increase in Objective Investigator Tolerability Parameters at week 4, 8, 12 compared to Baseline | 12 weeks
  The primary tolerability endpoint will be favorable analysis of the Investigator Tolerability Assessment of Erythema, Edema and Dryness. A change in scores or lack of significant change at week 4, week 8 and week 12 in comparison to Baseline indicates tolerability/safety of the test material. Four point scale with a lower score indicating a better outcome.
  Example for Erythema:
  0 = None No erythema of the treatment area, 1 = Mild Slight, but definite redness of the treatment area, 2 = Moderate Definite redness of the treatment area, 3 = Severe Marked redness of the treatment area
Incidence and severity of adverse events | 12 weeks
  The primary safety endpoint will be determined by the incidence and severity of adverse events in healthy subjects through-out the length of the study.

SECONDARY OUTCOMES:
Improvement in clinical efficacy of photodamage versus Baseline | 12 weeks
  The secondary efficacy endpoint will be the Investigator Clinical Grading using Modified Griffith's 10-point Scale. A change in scores at week 4, week 8 and week 12 in comparison to baseline indicates an improvement for the indicated parameter.
  Global facial photodamage will be assessed on each subject's face using a modified Griffiths' 10-point scale according to the following numerical definitions (half-point scores may be used as necessary to more accurately describe the skin condition): 0 = none (best possible condition); 1 to 3 = mild; 4 to 6 = moderate;7 to 9 = severe (worst possible condition). The lower the score equates to the best possible outcome.
Lack of Significant Increase in Objective Subject Tolerability Parameters at week 4, 8, 12 | 12 weeks
  The primary tolerability endpoint will be favorable analysis of the Subject Tolerability Assessment of Erythema, Edema and Dryness. A change in scores or lack of significant change at week 4, week 8 and week 12 in comparison to Baseline indicates tolerability/safety of the test material. Four point scale with a lower score indicating a better outcome.
  Example for Erythema: Erythema
  0=None No erythema of the treatment area,1=Mild Slight, but definite redness of the treatment area, 2=Moderate Definite redness of the treatment area, 3=Severe Marked redness of the treatment area

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Art of Skin MD, Solana Beach, California
  - About Skin, Greenwood Village, Colorado
  - Brian S. Biesman, M.D., Nashville, Tennessee

REFERENCES:
- [Derived] Hooper D, Tedaldi R, Iglesia S, Young MB, Kononov T, Zahr AS. Antioxidant Skincare Treatment for Hyperpigmented and Photodamaged Skin: Multi-Center, Open-Label, Cross-Seasonal Case Study. J Clin Aesthet Dermatol. 2023 Oct;16(10):31-38. PMID 37915337